CLINICAL TRIAL: NCT04986306
Title: The Validation of Sentinel Lymph Node Biopsy After Neo-adjuvant Chemotherapy in Breast Cancer Patients in National Cheng Kung University Hospital (NCKUH)
Brief Title: The Validation of Sentinel Lymph Node Biopsy After Neo-adjuvant Chemotherapy in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NCKUH SLNB
Record Dates: First submitted 2021-06-30; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer; Sentinel Lymph Node Biopsy; Neoadjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- clinical tumor stage 1-3 (cT1-3) and nodal stage 1 (cN1) breast cancer patients: Patients who will undergo neoadjuvant chemotherapy were asked to participate in this study. Informed consent will be given. Clip will be placed over the positive lymph node by surgeon which was proven by fine-needle aspiration cytology. After completion of neoadjuvant chemotherapy, surgery of the breast and the axilla was executed in the same session. Different surgeons performed the procedure.
  Interventions: Procedure: SLNB + ALND

INTERVENTIONS:
Procedure: SLNB + ALND — Patients who received neoadjuvant chemotherapy will undergo SLNB+ALND to evaluate the feasibility of SLNB

SUMMARY:
Neoadjuvant or primary systemic treatment is increasingly applied in the treatment of operable breast cancer. Down staging of the primary tumor is one of the important goals of neoadjuvant chemotherapy treatment (NCT), thereby permitting breast-conserving treatment without affecting the risk for a local relapse. Complete pathological response (pCR) rates after NCT vary across histological subtypes and can be more than 60% in HER2-positive disease with dual blockade therapy. Down staging of the axilla is also observed in patients initially presenting with metastatic lymph nodes. pCR rates in the axilla vary between 22% and 42% in reported series, again depending on tumor subtype. Omission of axillary lymph node dissection (ALND) can avoid the post-operative morbidity such as lymphedema in the short or long term follow-up.

Metastatic lymph node status is hard to be stated as a pCR in the axilla by using physical examination or imaging such as ultrasonography or tomography after complete NCT. Good response to the axilla lymph node causing the difficulty of tissue proof by using core needle biopsy, though the investigator knew that biopsy stands for the definite tool for the confirmation of the residual disease. One proposed method to decrease the false-negative rate (FNR) is clip placement in the positive node at initial diagnosis with confirmation of clipped node resection at surgery.

The correlation between the axillary lymph node identified on initial axillary ultrasound and the sentinel lymph nodes (SLNs) identified at surgery has not been fully evaluated. The concordance between percutaneous biopsy and the lymph node resected at the time of SLNB is not 100%. Sometimes, the initial node identified by ultrasound is not one of the SLNs. The impairment of the performance of SLNB might correlated to the alteration of lymphatic flow induced by tissue fibrosis or tumor deposits after NCT.

The investigator hypothesized that the clip placement at diagnosis of node-positive disease with removal of the clipped node during SLNB reduces the FNR of SLNB after NCT. Here, we evaluate how often the lymph node containing the clip placed at percutaneous biopsy before chemotherapy was found at surgery to be one of the SLNs, and how often it was found in the nodes retrieved at ALND. In addition, the investigator report the impact of identification of the clipped node within the SLNs on the FNR of SLNB.

DETAILED DESCRIPTION:
Aim 1: Identify the pathological result of SLN and ALN

Hypothesis:

The lymph node containing the clip placed at percutaneous biopsy before chemotherapy was found at surgery to be one of the SLNs

Method:

This study is a prospective study. 30 patients who will undergo neoadjuvant chemotherapy were asked to participate in this study. Informed consent will be given. Clip will be placed over the positive lymph node by surgeon which was proven by fine-needle aspiration cytology. After completion of neoadjuvant chemotherapy, surgery of the breast and the axilla was executed in the same session. Different surgeons performed the procedure.

The SLNB will be performed by dual tracer (blue dye plus indocyanine green or radioisotope). After remove the SLNs and ALN, detection of the clipped node will be identified under mammography-guided. The clipped lymph node will be marked separately. All of the lymph node will be sent to pathologist for final examination.

Aim 2: Check the feasibility of SLNB after neoadjuvant CT

Hypothesis:

SLNB is feasible after neoadjuvant CT under certain circumstances.

Method:

The primary endpoints used for statistical analysis were the success rate for identifying and selectively removing the clipped node and the correlation of the response observed in the clipped node on pathology with the ALND specimen. The identification rate of the clipped node was analyzed in all patients who underwent surgical removal of the clipped node. Correlation between the pathologic response observed in the clipped node and in the ALND specimen was estimated using false-negative rates, sensitivity, specificity, positive predictive value, negative predictive value, and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years.
* Female
* Primary breast cancer, not metastasis from other cancer.
* Histological subtypes: invasive ductal carcinoma.
* Clinical stage: cT1-3, cN1, cM0.
* Clip localization over at least one axillary lymph node.
* After neoadjuvant chemotherapy (NCT). The inclusion criteria and regimens of NCT are followed standard guildline of National Cheng Kung University Hospital.
* Complete response or partial response after NCT.
* Written inform consent.

Exclusion Criteria:

* Refuse to join the study.
* Unable to complete standard regimens of NCT.
* Metastasis in internal mammary nodes or other distant lymph nodes.
* Pregnancy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Groups will be formed of the breast cancer patients who meet the eligible criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The impact of clipped lymph node in patients who received SLNB and ALND following neoadjuvant chemotherapy | immediately after the surgery
  compare the location of clipped lymph node in SLNB or ALND

SECONDARY OUTCOMES:
Correlation of the pathologic response observed in the clipped node and SLNB | immediately after the surgery
  estimate the accuracy of SLNB by using false-negative rates, sensitivity, specificity, positive predictive value, negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Loh, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided